CLINICAL TRIAL: NCT05095285
Title: The Effect of Swaddling and Oropharyngeal Colostrum During Endotracheal Suctioning on Procedural Pain and Comfort in Premature Neonates.
Brief Title: Pain and Comfort During Endotracheal Suction in Premature Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Huriye Karadede, Research Assistant, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulAU
Record Dates: First submitted 2021-09-10; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Premature
Keywords: endotracheal suction; pain; comfort; swaddling; colostrum
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group (No Intervention): • In addition to incubator cover and nesting, no other non-pharmacological intervention was applied to the control group.
- The swaddling group (Experimental): •Babies in this group were wrapped with a white cheesecloth 2 minutes before ES in addition to incubator cover and nesting.
  Interventions: Other: Swaddling
- The oropharyngeal colostrum group (Experimental): • In addition to incubator cover and nesting, babies in this group were given 0.4 ml of colostrum with an insulin injector on the inside of the cheeks and on the tongue.
  Interventions: Other: Oropharyngeal colostrum

INTERVENTIONS:
Other: Swaddling — * Babies in this group were wrapped with a white cheesecloth 2 minutes before ES in addition to incubator cover and nesting.
  * Common procedure steps:
    * Legal representatives of the infants will sign an informed consent form.
    * İncubator cover and nesting
    * Endotracheal suction(ES) was performed in the supine position.
    * ES was done at the time of care the baby needed.
    * No painful procedure was applied until 2 hours before ES and 15 minutes after ES.
    * Aspiration was performed sterile at 80 mmHg pressure.
    * A second nurse assisted in the suction process and the procedure took no more than 15 seconds.
    * The amount of oxygen taken by the baby was increased by 10% 30 seconds before the suction procedure and returned to its original value 60 seconds after the procedure.
    * Beginning 3 minutes before the ES procedure, during the procedure and until 15 minutes after the procedure, the infants' behaviors and bedside monitor indicators were video recorded.
  Arms: The swaddling group
Other: Oropharyngeal colostrum — * Common procedure steps
  * In addition to incubator cover and nesting, babies in this group were given 0.4 ml of colostrum with an insulin injector on the inside of the cheeks and on the tongue.
  Arms: The oropharyngeal colostrum group

SUMMARY:
Most of the preterm babies in neonatal units are followed up with invasive mechanical ventilation support. For this reason, endotracheal suction is needed repeatedly in preterm babies in order to open the airway obstruction caused by secretions and to maintain the airway patency. Endotracheal aspiration, which is one of the invasive procedures in which pain is felt most in newborns, is performed by nurses.

Endotracheal suction, which causes pain and discomfort in intensive care units, negatively affects the comfort of patients. Studies emphasize that comfort is an indicator of pain and stress, and the comfort scale is also used in pain and distress assessments.

Effective pain management and the development of pain-related care standards to reduce pain in preterm newborn infants improve clinical and neurodevelopmental outcomes. For this reason, it is necessary to reduce the pain that has an effect on the development of preterm babies.

In pediatric nursing, studies on non-pharmacological methods have increased in recent years in order to increase the comfort of infants and reduce pain and stress, especially during painful and stressful procedures in infants followed in neonatal intensive care units. When the literature is examined, there are few studies measuring the effectiveness of non-pharmacological methods used in reducing pain due to endotracheal suction. There are differences in the effectiveness of the methods applied in the existing studies. Therefore, more observation, research and scientific studies by neonatal nurses are needed to reduce the pain associated with endotracheal suction in preterm newborns.

In this study, swaddling and oropharyngeal colostrum, which are two non-pharmacological methods, will be applied during endotracheal suction to preterm newborns receiving invasive mechanical ventilation support. This experimental study was planned to determine the effect of these two non-pharmacological methods on procedural pain and comfort and to contribute to evidence-based nursing practices.

DETAILED DESCRIPTION:
The study was conducted experimentally in randomized controlled trials to determine the effect of two non-pharmacological methods, swaddling and oropharyngeal colostrum on procedural pain and comfort during endotracheal suction (ES) in premature neonates. The population of the study was intubated premature neonates hospitalized in NICU in two foundation university hospitals between July 2019 and October 2020. The study sample consisted of 48 babies who met the sample selection criteria. Descriptive Characteristics Form, Premature Infant Intervention Follow-up Form, Premature Infant Pain Profile-Revised (PIPP-R) and Newborn Comfort Behavior Scale (COMFORTneo) were used in data collection.

Two minutes before the ES procedure, babies were swaddled or 0.4 ml of oropharyngeal colostrum was given, depending on the group in which they were involved. Physiological parameters (heart rate, respiration, saturation) of the babies were recorded before, during and after the procedure, and PIPP-R and COMFORTneo scores were given by two observers by video recording.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age of the baby is 26-36 weeks according to the mother's last menstrual period
* Baby's postnatal 0-5. be between days
* Receiving invasive mechanical ventilation support
* No analgesic, opioid and sedative pain relievers were administered in the 4 hours before the procedure.
* It has been 2 hours since the last painful attempt.
* Parental consent of the premature baby.
* Applying endotracheal suction at most 2 times since birth

Exclusion Criteria:

* Presence of congenital anomaly
* Having a history of convulsions
* Any extremity fracture/dislocation that will prevent wrapping
* Having a pneumothorax tube

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate | Baby's heart rate will monitored during 20 minutes since it will start the camera record. (Heart rates will be evaluated at baseline, 2 minutes, during endotracheal suction(ES), immediately after ES, 5 minutes, 10 minutes, 15 minutes later.)
  Heart rate will be monitored
Change in Oxygen Saturation | Baby's oxygen saturation will monitored during 20 minutes since it will start the camera record. (Oxygen Saturation will be evaluated at baseline, 2 minutes, during endotracheal suction(ES), immediately after ES, 5 minutes, 10 minutes, 15 minutes later.)
  Oxygen saturation will be monitored
Change in pain score | Baby's pain score will be evaluated during 20 minutes since it will start the camera record. (Pain score will be evaluated at baseline, 2 minutes, during endotracheal suction(ES), immediately after ES, 5 minutes, 10 minutes, 15 minutes later.)
  Pain score will be evaluated with Premature Infant Pain Profile-Revised (PIPP-R).
Change in comfort score | Baby's comfort score will be evaluated during 20 minutes since it will start the camera record. (Comfort score will be evaluated at baseline, 2 minutes, during endotracheal suction(ES), immediately after ES, 5 minutes, 10 minutes, 15 minutes later.)
  Comfort score will be evaluated with Newborn Comfort Behavior Scale (COMFORTneo)

SECONDARY OUTCOMES:
Change in Respiratory Rate | Baby's respiratory rate will be monitored during 20 minutes since it will start the camera record. (Respiratory Rate will be evaluated at baseline, 2 minutes, during endotracheal suction(ES), immediately after ES; 5, 10 and 15 minutes later.)
  Respiratory Rate will be monitored
Change in Body temperature | Baby's body temperature will be measurement during 20 minutes since it will start the camera record. (Body temperature will be measurement at baseline, 2 minutes, during endotracheal suction(ES), immediately after ES; 5, 10 and 15 minutes later.)
  Body temperature will be measurement
Change in blood pressure | Baby's blood pressure will be monitored during 20 minutes since it will start the camera record. (Blood pressure will be monitored at baseline, 2 minutes, during endotracheal suction(ES), immediately after ES, 5 minutes, 10 minutes, 15 minutes later.)
  Blood pressure will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Mutlu, Ass. Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Desai S, Nanavati RN, Nathani R, Kabra N. Effect of Expressed Breast Milk versus Swaddling versus Oral Sucrose Administration on Pain Associated with Suctioning in Preterm Neonates on Assisted Ventilation: A Randomized Controlled Trial. Indian J Palliat Care. 2017 Oct-Dec;23(4):372-378. doi: 10.4103/IJPC.IJPC_84_17. PMID 29123341
- [Result] Taplak AS, Bayat M. Comparison the Effect of Breast Milk Smell, White Noise and Facilitated Tucking Applied to Turkish Preterm Infants During Endotracheal Suctioning on Pain and Physiological Parameters. J Pediatr Nurs. 2021 Jan-Feb;56:e19-e26. doi: 10.1016/j.pedn.2020.07.001. Epub 2020 Jul 18. PMID 32690406
- [Result] Stevens BJ, Gibbins S, Yamada J, Dionne K, Lee G, Johnston C, Taddio A. The premature infant pain profile-revised (PIPP-R): initial validation and feasibility. Clin J Pain. 2014 Mar;30(3):238-43. doi: 10.1097/AJP.0b013e3182906aed. PMID 24503979
- [Result] Taplak AS, Bayat M. Psychometric Testing of the Turkish Version of the Premature Infant Pain Profile Revised-PIPP-R. J Pediatr Nurs. 2019 Sep-Oct;48:e49-e55. doi: 10.1016/j.pedn.2019.06.007. Epub 2019 Jun 19. PMID 31229348
- [Result] Apaydin Cirik V, Efe E. The effect of expressed breast milk, swaddling and facilitated tucking methods in reducing the pain caused by orogastric tube insertion in preterm infants: A randomized controlled trial. Int J Nurs Stud. 2020 Apr;104:103532. doi: 10.1016/j.ijnurstu.2020.103532. Epub 2020 Jan 24. PMID 32062050
- [Result] Kucuk Alemdar D, Guducu TufekcI F. Effects of maternal heart sounds on pain and comfort during aspiration in preterm infants. Jpn J Nurs Sci. 2018 Oct;15(4):330-339. doi: 10.1111/jjns.12202. Epub 2018 Jan 17. PMID 29345047
- [Result] Cardoso JM, Kusahara DM, Guinsburg R, Pedreira ML. Randomized crossover trial of endotracheal tube suctioning systems use in newborns. Nurs Crit Care. 2017 Sep;22(5):276-283. doi: 10.1111/nicc.12170. Epub 2015 Mar 16. PMID 25779636